CLINICAL TRIAL: NCT04688736
Title: A Prospective, Randomized, Double-blind Controlled Trial of Chlorpheniramine Pretransfusion Medication for Allergic Transfusion Reactions
Brief Title: Efficacy of Placebo Versus Chlorpheniramine for the Prevention of Allergic Transfusion Reactions.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IIT2020032
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-03

CONDITIONS: Allergic Transfusion Reaction
Keywords: pretransfusion medication; Chlorpheniramine; blood transfusion; allergic transfusion reaction
MeSH Terms: interventions — Chlorpheniramine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither patients nor medical staff, including physicians and nurses participating in this study, will know the group assignment after allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Experimental): Each recruited subject will oral 8mg placebo 20 minutes before blood transfusion.
  Interventions: Drug: Placebo
- Chlorpheniramine (Active Comparator): Each recruited subject will oral 8mg chlorpheniramine 20 minutes before blood transfusion.
  Interventions: Drug: Chlorpheniramine

INTERVENTIONS:
Drug: Placebo — The tablet resembles chlorpheniramine but has no therapeutic value.
  Arms: Placebo
Drug: Chlorpheniramine — An antihistamine that reduces the natural chemical histamine in the body.
  Arms: Chlorpheniramine

SUMMARY:
This is a prospective, randomized, double-blind controlled trial to evaluate the efficacy of placebo versus chlorpheniramine for the prevention of allergic transfusion reactions.

ELIGIBILITY:
Inclusion Criteria:

* 18~65 years old.
* Subject is diagnosed with hematological disorder and requires blood product (i.e. suspended red blood cells, apheresis platelets, fresh frozen plasma) transfusions.
* Subject can fully understand and voluntarily sign informed consent forms.

Exclusion Criteria:

* Subject with a history of allergic diseases.
* Subject experienced at least 1 moderate/severe or 2 mild allergic reactions in the past.
* Subject received glucocorticoid or allergy drugs within 24 hours before blood transfusion.
* Subject transfused with washed RBC.
* Received allo-HSCT transplantation before.
* Subject with heart failure.
* Subject suffered from sequelae of cardiovascular or cerebrovascular diseases.
* Pregnant or nursing women.
* Inability to understand or to follow study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6642 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
The rate of allergic-transfusion reactions | within 4 hours from the start of the transfusion

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Zhoukou Central Hospital, Zhoukou, Henan
  - The Second Affilated Hospital of Shandong First Medical University, Tai’an, Shandong
  - Regenerative Medicine Center, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No